CLINICAL TRIAL: NCT05005793
Title: Effect of Alkali Therapy on Vascular and Graft Function in Kidney Transplant
Brief Title: Effect of Alkali Therapy on Vascular and Graft Function in Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-3447; R01DK130255 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-08-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Acidosis; Kidney Transplant; Complications; Vascular Diseases
MeSH Terms: conditions — Acidosis; Vascular Diseases | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): Oral sodium bicarbonate at a dose of 0.5 mEq/kg-lean body weight/day
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): Oral placebo at a dose of 0.5 mEq/kg-lean body weight/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — Oral sodium bicarbonate at 0.5 mEq/kg-lean body weight/day
  Arms: Sodium bicarbonate
Drug: Placebo — Placebo at 0.5 mEq/kg-lean body weight/day
  Arms: Placebo

SUMMARY:
Lower serum bicarbonate levels, even within the normal laboratory range, in kidney transplant recipients (KTRs) are associated with an increased risk of graft loss, cardiovascular events and mortality. Because acid retention is common in KTRs, it is plausible that alkali therapy in KTRs may also result in improved vascular and graft function. The investigators will perform a randomized, double-blinded, placebo-controlled, 12 month study in 120 KTRs to examine the effect of sodium bicarbonate therapy on surrogate markers of CVD and graft function. The overall hypothesis is that treatment with bicarbonate will improve indicators of vascular and graft function in KTRs by decreasing complement activation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Serum bicarbonate 16-24 mEq/L on 2 separate measurements (at least 1 day apart)
* Kidney transplant received 1 year prior to randomization
* eGFR ≥ 45 ml/min/1.73m2 by CKD-EPI equation
* Blood pressure <130/80 mm Hg prior to randomization
* BMI < 40 kg/m2 (FMD measurements can be inaccurate in severely obese patients).
* Able to provide consent
* Immunosuppression regimen consisting of tacrolimus, mycophenolate mofetil and prednisone (95% of patients at University of Colorado are on this regimen)
* Stable immunosuppression regimen for at least three months prior to randomization
* Stable anti-hypertensive regimen for at least one month prior to randomization
* Not taking medications that interact with agents administered during experimental sessions (e.g. sildenafil interacts with nitroglycerin).

Exclusion Criteria:

* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Use of chronic daily oral alkali within the last 3 months (including sodium bicarbonate, calcium carbonate or baking soda)
* Uncontrolled hypertension
* Serum potassium < 3.3 or ≥ 5.5 mEq/L at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known EF ≤30%, or hospital admission for heart failure within the past 3 months
* Nephrotic range proteinuria (urine complement activation fragment measurements may not be accurate with severe proteinuria)
* Factors judged to limit adherence to interventions
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Chronic use of supplemental oxygen
* Use of anticoagulants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brachial artery flow mediated dilation at 12 months | Baseline and 12 months
  Brachial artery FMD will be determined using high-resolution ultrasonographyECG-gated end-diastolic ultrasound images and Doppler flow of the brachial artery will be acquired during baseline and FMD conditions. For FMD, reactive hyperemia will be produced by inflating a pediatric BP cuff around the forearm to 250 mmHg for 5 minutes followed by rapid deflation.

SECONDARY OUTCOMES:
Change in Large elastic artery stiffness and compliance at 12 months | Baseline and 12 months
  transcutaneous custom tonometers (Noninvasive hemodynamics Workstation, Cardiovascular Engineering Inc., Norwood, MA) will be positioned at the aorta and femoral artery to measure aortic pulse wave velocity.
Change in Tubular atrophy at 12 months | Baseline and 12 months
  Kidney transplant biopsies will be performed. Morphometric analysis will be performed using trichrome and Sirius Red to determine tubular atrophy. All imaging will be done using an Aperio scanner.
Change in participant plasma and urine complement activation fragment levels at 12 months | Baseline and 12 months
  Complement activation fragments (Ba, C4a, C3a, C5a, sC5b-9) will be measured at the University of Colorado Exsera Biolab located on the Anschutz Medical Campus.
Change in interstitial fibrosis at 12 months | Baseline and 12 months.
  Kidney transplant biopsies will be performed. Morphometric analysis will be performed using trichrome and Sirius Red to determine interstitial fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD MPH, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the study, data, which has been stripped of all personal identification information and coded with a number, will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of this study will be made generally available by publication and journal articles submitted to PubMed Central in compliance with NIH access guidelines.